CLINICAL TRIAL: NCT05803239
Title: The Diagnostic Yield and Safety of Endobronchial Ultrasound-guided Mediastinal Cryobiopsy Via a Tunnel in Mediastinal Lymphadenopathy
Brief Title: Study on Endobronchial Ultrasound-guided Transbronchial Mediastinal Cryobiopsy Via a Tunnel in the Diagnosis of Mediastinal Lymphadenopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-NHLHCRF-LX-01-0201-03
Record Dates: First submitted 2023-03-14; First posted 2023-04-07 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-05

CONDITIONS: Mediastinal Lymphadenopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EBUS-TBMC via a tunnel first group (Experimental): After completing the routine bronchoscopy examination, under the EBUS guidance, combined with the results of chest CT to determine the location of puncture. Then, a disposable puncture dilation catheter (BroncTru AK-91-55; Broncus Inc., Hangzhou, China) was inserted through the working channel of the ultrasound bronchoscope and built a tunnel between the airway wall and targeted lymph node. The 1.1-mm cryoprobe (Erbe 20402-401; ERBE, Tübingen, Germany) was inserted into the target lymph node through the tunnel under direct EBUS monitoring, and the distance between the tip of the cryoprobe and the border of the target lymph node was measured using EBUS. After confirming that the distance was >5 mm, the probe was cooled with liquid carbon dioxide for 5-9 seconds and freezing 3 times to obtain 3 pieces of sample. At the end of TBMC via a tunnel, EBUS-TBNA is performed in the same lymph node, and the tissue is aspirated repeatedly for 5 strokes (one stroke is 30 round trips).
  Interventions: Procedure: EBUS-TBNA; Procedure: EBUS-TBMC via a tunnel
- EBUS-TBNA first group (Experimental): Completion of routine bronchoscopy, determination of the puncture position under EBUS guidance, combined with the results of chest CT, and application of the EBUS-TBNA needle to repeatedly aspirate the tissue for 5 strokes (one stroke is 30 round trips ). At the end of the puncture, EBUS-TBMC via a tunnel was then performed with a freezing time of 5-9 seconds (1.1-mm cryoprobe), and frozen 3 times to obtain 3 pieces of samples.
  Interventions: Procedure: EBUS-TBNA; Procedure: EBUS-TBMC via a tunnel

INTERVENTIONS:
Procedure: EBUS-TBNA — Participants with lymphadenopathy would receive EBUS-TBNA attempts to conduct diagnoses.
Procedure: EBUS-TBMC via a tunnel — Participants with lymphadenopathy would receive EBUS-TBMC via a tunnel attempts to conduct diagnoses.

SUMMARY:
The goal of this clinical trial is to clear the diagnostic yield and safety of endobronchial ultrasound-guided transbronchial mediastinal cryobiopsy (TBMC) via a tunnel. The main questions it aims to answer are:

Does EBUS-TBMC via a tunnel have a superior diagnostic yield to EBUS-transbronchial needle aspiration (TBNA)? When EBUS-TBMC via a tunnel could be performed as a first-line diagnostic tool in patients with mediastinal and/or hilar lymphadenopathy?

Researchers will compare EBUS-TBMC via a tunnel to EBUS-TBNA to see if EBUS-TBMC via a tunnel has a superior of diagnostic yield with a well-tolerance.

Participants will:

Recieve EBUS-TBMC via a tunnel and EBUS-TBNA in a predefined sequence. Recieve chest CT examination and follow-up for 7 days after procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one mediastinal and/or hilar lymphadenopathy (≥1cm in the short axis) in the absence of a known or suspected primary lung cancer, requiring diagnostic bronchoscopy.
* The selected patients should complete the routine examination of EBUS-TBNA/EBUS-TBMC via a tunnel before operation, such as blood routine examination, coagulation function, electrocardiogram, chest CT, etc.
* There was no contraindication of puncture and cryobiopsy.
* Fully informed of the purpose and method of the study, agreed to participate in the study, and signed the informed consent form.

Exclusion Criteria:

* The lesion is a mediastinal cyst or abscess.
* The patient is allergic to lidocaine and midazolam.
* The site to be biopsied has a high risk of bleeding detected by Doppler and/or contrast CT such as bronchial artery penetration or suspected lung metastasis of renal cancer.
* Unstable angina pectoris, congestive heart failure, severe bronchial asthma
* The patient did not agree to participate in this study
* Participation in other studies within three months without withdrawal or termination will affect the observation of this study
* The researcher believes that there is any person who is not suitable for the selection

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2023-02-18 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield | 6 months after the biopsy
  The proportion of all individuals undergoing the diagnostic procedure under evaluation in whom a specific diagnosis was established. All the final diagnosis in this trial were established by the treating clinician and verified by an independent diagnosis verification panel which included three pulmonary and critical care medicine physicians, one radiologist, and one pathologist.

SECONDARY OUTCOMES:
Diagnostic sensitivity | 6 months after biopsy.
  The proportion of individuals who truly had the disease and tested positive.
Incidence rate of adverse events | 7 days after the biopsy
  Symptoms and signs
Size of specimen | during the procedure
  measurement
Specimen quality | during the procedure
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gang Hou, MD, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No